CLINICAL TRIAL: NCT03096093
Title: A Phase I Clinical Study to Determine the Optimal Dose for the Safe Immune Restoration and Immune Response of Allogeneic Cell Immunotherapy (ACIT-1) in Adult Cancer Patients
Brief Title: Investigation of a Therapeutic Vaccine (ACIT-1) in Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Vaccines Limited (Industry)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); The Clatterbridge Cancer Centre NHS Foundation Trust (Other); University of Liverpool (Other); Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government); Cancer Vaccines Charitable Trust (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACIT-1-1001; 2012-005426-30 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Neoplasms
Keywords: Pancreatic; Late stage cancer; Immunotherapy; Phase I; Vaccination
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immunotherapy - pancreatic cancer (Experimental): Intradermal injection of ACIT-1 cellular immunotherapy, a total of 2 doses, 4 weeks apart of either 10e5, 10e6, 10e7 or 3x10e7 cells. For patients with pancreatic or haematological cancer. Treatment will run concurrently with standard chemotherapy.
  Interventions: Biological: ACIT-1
- Immunotherapy - other late stage cancers (Experimental): Intradermal injection of ACIT-1 cellular immunotherapy, a total of 2 doses, 4 weeks apart of either 10e5, 10e6, 10e7 or 3x10e7 cells. For patients with other late stage cancers, not receiving any other standard treatment.
  Interventions: Biological: ACIT-1

INTERVENTIONS:
Biological: ACIT-1 — Cell suspension

SUMMARY:
This study evaluates four different doses of ACIT-1 for safety and for the ability to raise effective anti-cancer immune responses in patients with pancreatic and other cancers. Approximately half of the patients will have pancreatic cancer and the other half will have other cancers.

DETAILED DESCRIPTION:
The immune system has an important role in helping prevent cancer by destroying early cancer cells. When cancer does develop antigen-specific immune (T) cells are still present in the blood but are either not responding or are not effective. Vaccines stimulate these T cells to respond and kill cancer cells.

ACIT-1 is designed to stimulate tumour antigen-specific T cells to respond and kill cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* Life-expectancy of 3 months or greater
* Aged 18 years or above
* Willing and able to give written informed consent for participation in the study
* Eastern Cooperative Oncology Group performance status of 0,1,2.
* Absolute neutrophil count of ≥ 1 x 10e12/m3
* Platelet count of at least 70 x 10e12/m3
* Total bilirubin < 1.5x upper limit of normal; and aspartate transaminase/alanine transaminase (AST/ALT) < 5x upper limit of normal
* Creatinine < 1.5x upper limit of normal and/or glomerular filtration rate (GFR) > 40ml/min
* Female patients of child bearing potential and male patients whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Normal ECG measurements
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner (GP) and consultant, if appropriate, to be notified of participation in the study, and for the GP and/or the National Cancer Registry to be contacted during follow up after the end of treatment.

Exclusion Criteria:

* Concurrent use of immunosuppressive drugs, in particular systemic steroid therapy, above a threshold of 10mg per day prednisolone equivalent
* Evidence of active infection e.g. Hepatitis B, Hepatitis C, HIV or syphilis
* Chemotherapy, radiotherapy or biological therapy within 28 days of treatment with the exception of standard of care chemotherapy for pancreatic and haematological cancer patients
* Participation in another investigational medicinal product trial within 28 days of treatment
* Other vaccination within previous 4 weeks
* Antibody treatment within previous 3 months
* Major surgery within the 14 days preceding the screening visit
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Allogeneic graft transplantation recipient
* Active systemic autoimmune and allergic disease
* Pregnant or lactating females
* Significant renal or hepatic impairment as defined by the following: Serum creatinine ≥ 1.5 x upper limit of normal and/or GFR ≤ 40 ml/min. Total bilirubin ≥ 1.5 x upper limit of normal; and AST/ALT ≥ 5 x upper limit of normal
* Life threatening illness unrelated to the patient's cancer
* Previous history of serious adverse allergic reaction to any medication
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity | From start of treatment to 20 weeks.
  Toxicity based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.

SECONDARY OUTCOMES:
Clinical benefit | From start of treatment up to 14 months.
  Survival time

OTHER OUTCOMES:
Immune responses | Baseline, weeks 4, 8 and 20
  Changes in tumour antigen specific immune responses in the blood compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Palmer, MBChB PhD, Principal Investigator — Clatterbridge Cancer Centre
Locations (2):
- United Kingdom (2):
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral

IPD SHARING:
Plan to Share IPD: No